CLINICAL TRIAL: NCT03096678
Title: Morphological and Functional Changes, Risk Stratification and Prognosis of Patients With Compete Left Bundle Branch Block
Brief Title: Prognosis of Patients With Compete Left Bundle Branch Block
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Collaborators: Beijing Anzhen Hospital (Other); China-Japan Friendship Hospital (Other); Peking Union Medical College Hospital (Other); Xuanwu Hospital, Beijing (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Minjie Lu, Principal Investigator, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: LBBB001
Record Dates: First submitted 2017-03-25; First posted 2017-03-30 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Bundle-Branch Block, Left; Cardiac Failure; ICD/Pacemaker Implantation; Cardiovascular Magnetic Resonance Imaging
Keywords: Left Bundle Branch Block; Regional/Globle cardiac function; Mechanical asynchrony; Cardiovascular Magnetic Resonance; Outcome; Cardiovascular events
MeSH Terms: conditions — Bundle-Branch Block; Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LBBB without LV dysfunction: LVEDD>55mm or LVEF<55%
  Interventions: Diagnostic Test: Cardiac Magnetic Resonance Imaging
- LBBB with LV dysfunction: LVEDD<55mm and LVEF>55%
  Interventions: Diagnostic Test: Cardiac Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: Cardiac Magnetic Resonance Imaging — Using a comprehensive MR study (Function, LGE, Tissue Characterization, Strain, T1/T2 mapping) to predict the outcome of LBBB with different cardiac function.

SUMMARY:
The investigators sought to evaluate the morphological and functional changes, risk stratification and prognosis of patients of participants with compete left bundle branch block (CLBBB).

The conduction of this study was largely due to the increased clinical requirement, which reflected the increased awareness among physicians of heart failure due to asynchronous cardiac function caused by CLBBB. The investigators also aim to figure out the time point or CMR parameters for cardiac resynchronization therapy in patients with CLBBB.

DETAILED DESCRIPTION:
The effect of cardiac resynchronization therapy (CRT) for heart failure patients was heterogeneous. Candidate selection was important before intervention. The underlying mechanical dyssynchrony of left ventricular bundle branch block was insufficiently descripted. Earlier study of investigators found novel imaging methods such as cardiovascular magnetic resonance imaging including T1 Mapping and feature tracking imaging can provide more detailed information about regional and global LV function in patients. While the role of new cardiac MR imaging techniques in predicting CRT responses, especially in LBBB patients, is still insufficient. Z Chen et al used T1 mapping technique to quantitatively assess the diffuse fibrosis burden of myocardial in heart failure patients. But they found focal fibrosis burden, not diffuse burden, is associated with a poor response to CRT. Other cardiac MR imaging parameters also showed potential predictors of CRT, such as 16 segment time-to-maximum radial wall thickness , scar locations and RV septal lead placement.In this study cardiovascular magnetic resonance imaging (including T1 Mapping combined with feature tracking imaging ) will be applied to follow up LV function in LBBB patients (with or without intervention) in 10 years to find out prognostic predictors and time point or CMR parameters for cardiac resynchronization therapy in patients with CLBBB.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years or older and able and willing to consent.
* The patient should present a complete left bundle branch block (LBBB) with QRS duration of >120ms
* The patients should be in NYHA functional class I, II or III.

Exclusion Criteria:

* No informed consent
* Permanent atrial fibrillation, flutter or tachycardia (>100 bpm).
* Right bundle branch block
* Recent myocardial infarction, within 40 days prior to enrolment.
* Subject underwent coronary artery bypass graft (CABG) or valve surgery, within 90 days.
* Implanted with a LV assist device (LVAD), or has reasonable probability (per investigator's discretion) of receiving a LVAD in the next year.
* Severe aortic stenosis (with a valve area of <1.0 cm2 or significant valve disease expected to be operated on within study period).
* Complex and uncorrected congenital heart disease.
* Claustrophobia or devices

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: subjects with complete left bundle branch block
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause death | 10 years
Cardiovascular death | 10 years
Heart Transplantation | 10 years

SECONDARY OUTCOMES:
ICD Implantation | 10 years
Pacemaker Implantation | 10 years
Myocardial Infarction | 10 years
Hospitalization due to heart failure | 10 years
Stroke | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Minjie Lu, MD,PhD, Study Chair — Fuwai Hospital, State Key Laboratory of Cardiovascular Disease, Fuwai Hospital, National Center for Cardiovascular Diseases, Chinese Academy of Medical, Sciences and Peking Union Medical College
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Flowers NC. Left bundle branch block: a continuously evolving concept. J Am Coll Cardiol. 1987 Mar;9(3):684-97. doi: 10.1016/s0735-1097(87)80065-7. PMID 2950157
- [Background] Ansalone G, Giannantoni P, Ricci R, Trambaiolo P, Fedele F, Santini M. Biventricular pacing in heart failure: back to basics in the pathophysiology of left bundle branch block to reduce the number of nonresponders. Am J Cardiol. 2003 May 8;91(9A):55F-61F. doi: 10.1016/s0002-9149(02)03339-8. PMID 12729851
- [Background] Marsan NA, Westenberg JJ, Ypenburg C, van Bommel RJ, Roes S, Delgado V, Tops LF, van der Geest RJ, Boersma E, de Roos A, Schalij MJ, Bax JJ. Magnetic resonance imaging and response to cardiac resynchronization therapy: relative merits of left ventricular dyssynchrony and scar tissue. Eur Heart J. 2009 Oct;30(19):2360-7. doi: 10.1093/eurheartj/ehp280. Epub 2009 Jul 4. PMID 19578165
- [Background] Sohal M, Shetty A, Duckett S, Chen Z, Sammut E, Amraoui S, Carr-White G, Razavi R, Rinaldi CA. Noninvasive assessment of LV contraction patterns using CMR to identify responders to CRT. JACC Cardiovasc Imaging. 2013 Aug;6(8):864-73. doi: 10.1016/j.jcmg.2012.11.019. Epub 2013 Jun 2. PMID 23735442
- [Background] Kellman P, Hansen MS. T1-mapping in the heart: accuracy and precision. J Cardiovasc Magn Reson. 2014 Jan 4;16(1):2. doi: 10.1186/1532-429X-16-2. PMID 24387626
- [Background] Ambale-Venkatesh B, Lima JA. Cardiac MRI: a central prognostic tool in myocardial fibrosis. Nat Rev Cardiol. 2015 Jan;12(1):18-29. doi: 10.1038/nrcardio.2014.159. Epub 2014 Oct 28. PMID 25348690
- [Background] Risum N, Tayal B, Hansen TF, Bruun NE, Jensen MT, Lauridsen TK, Saba S, Kisslo J, Gorcsan J 3rd, Sogaard P. Identification of Typical Left Bundle Branch Block Contraction by Strain Echocardiography Is Additive to Electrocardiography in Prediction of Long-Term Outcome After Cardiac Resynchronization Therapy. J Am Coll Cardiol. 2015 Aug 11;66(6):631-41. doi: 10.1016/j.jacc.2015.06.020. PMID 26248989
- [Background] Aurich M, Keller M, Greiner S, Steen H, Aus dem Siepen F, Riffel J, Katus HA, Buss SJ, Mereles D. Left ventricular mechanics assessed by two-dimensional echocardiography and cardiac magnetic resonance imaging: comparison of high-resolution speckle tracking and feature tracking. Eur Heart J Cardiovasc Imaging. 2016 Dec;17(12):1370-1378. doi: 10.1093/ehjci/jew042. Epub 2016 Mar 24. PMID 27013249
- [Background] Bogarapu S, Puchalski MD, Everitt MD, Williams RV, Weng HY, Menon SC. Novel Cardiac Magnetic Resonance Feature Tracking (CMR-FT) Analysis for Detection of Myocardial Fibrosis in Pediatric Hypertrophic Cardiomyopathy. Pediatr Cardiol. 2016 Apr;37(4):663-73. doi: 10.1007/s00246-015-1329-8. Epub 2016 Jan 30. PMID 26833321
- [Background] Puntmann VO, Carr-White G, Jabbour A, Yu CY, Gebker R, Kelle S, Hinojar R, Doltra A, Varma N, Child N, Rogers T, Suna G, Arroyo Ucar E, Goodman B, Khan S, Dabir D, Herrmann E, Zeiher AM, Nagel E; International T1 Multicentre CMR Outcome Study. T1-Mapping and Outcome in Nonischemic Cardiomyopathy: All-Cause Mortality and Heart Failure. JACC Cardiovasc Imaging. 2016 Jan;9(1):40-50. doi: 10.1016/j.jcmg.2015.12.001. PMID 26762873
- [Background] Taylor AJ, Salerno M, Dharmakumar R, Jerosch-Herold M. T1 Mapping: Basic Techniques and Clinical Applications. JACC Cardiovasc Imaging. 2016 Jan;9(1):67-81. doi: 10.1016/j.jcmg.2015.11.005. PMID 26762877
- [Background] van der Graaf AW, Bhagirath P, Scheffer MG, de Medina RR, Gotte MJ. MR feature tracking in patients with MRI-conditional pacing systems: The impact of pacing. J Magn Reson Imaging. 2016 Oct;44(4):964-71. doi: 10.1002/jmri.25229. Epub 2016 Mar 17. PMID 26990922
- [Background] Witt CM, Wu G, Yang D, Hodge DO, Roger VL, Cha YM. Outcomes With Left Bundle Branch Block and Mildly to Moderately Reduced Left Ventricular Function. JACC Heart Fail. 2016 Nov;4(11):897-903. doi: 10.1016/j.jchf.2016.07.002. Epub 2016 Sep 7. PMID 27614941
- [Background] Cerit L. Prediction of Readmission for Congestive Heart Failure With or Without Left Bundle Branch Block. Am J Cardiol. 2017 Jul 15;120(2):337. doi: 10.1016/j.amjcard.2017.01.010. Epub 2017 Feb 2. No abstract available. PMID 28233534
- [Background] Erne P, Iglesias JF, Urban P, Eberli FR, Rickli H, Simon R, Fischer TA, Radovanovic D. Left bundle-branch block in patients with acute myocardial infarction: Presentation, treatment, and trends in outcome from 1997 to 2016 in routine clinical practice. Am Heart J. 2017 Feb;184:106-113. doi: 10.1016/j.ahj.2016.11.003. Epub 2016 Nov 10. PMID 28224924
- [Background] Kawji MM, Glancy DL. Hypotension and Left Bundle Branch Block. Am J Cardiol. 2017 Apr 15;119(8):1292-1293. doi: 10.1016/j.amjcard.2016.11.070. Epub 2017 Jan 25. PMID 28258731
- [Result] Lu M, Zhao S, Jiang S, Yin G, Wang C, Zhang Y, Liu Q, Cheng H, Ma N, Zhao T, Chen X, Huang J, Zou Y, Song L, He Z, An J, Renate J, Xue H, Shah S. Fat deposition in dilated cardiomyopathy assessed by CMR. JACC Cardiovasc Imaging. 2013 Aug;6(8):889-98. doi: 10.1016/j.jcmg.2013.04.010. Epub 2013 Jul 10. PMID 23850250
- [Result] Lu M, Zhao S, Yin G, Jiang S, Zhao T, Chen X, Tian L, Zhang Y, Wei Y, Liu Q, He Z, Xue H, An J, Shah S. T1 mapping for detection of left ventricular myocardial fibrosis in hypertrophic cardiomyopathy: a preliminary study. Eur J Radiol. 2013 May;82(5):e225-31. doi: 10.1016/j.ejrad.2012.12.014. Epub 2013 Jan 17. PMID 23333530
- [Result] Lu M, Du H, Gao Z, Song L, Cheng H, Zhang Y, Yin G, Chen X, Ling J, Jiang Y, Wang H, Li J, Huang J, He Z, Zhao S. Predictors of Outcome After Alcohol Septal Ablation for Hypertrophic Obstructive Cardiomyopathy: An Echocardiography and Cardiovascular Magnetic Resonance Imaging Study. Circ Cardiovasc Interv. 2016 Mar;9(3):e002675. doi: 10.1161/CIRCINTERVENTIONS.115.002675. PMID 26884612